CLINICAL TRIAL: NCT00323453
Title: Rate of Surgical Wound Infection After Open Appendectomy Using the Alexis Wound Retractor
Brief Title: Wound Infection Alexis Wound Retractor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-06
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Appendicitis
Keywords: Appendectomy; Surgery; Infection
MeSH Terms: conditions — Appendicitis; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm (Experimental): The experimental arm will undergo open appendectomy utilizing the Alexis® retractor (wound protection device utilized intraoperatively), followed by standardized wound closure.
  Interventions: Device: Open appendectomy using Alexis Wound Retractor followed by standardized wound closure
- Control Arm (Placebo Comparator): Open appendectomy and standardized wound closure
  Interventions: Procedure: Open appendectomy with standardized wound closure

INTERVENTIONS:
Device: Open appendectomy using Alexis Wound Retractor followed by standardized wound closure — The control arm subjects will undergo open appendectomy and standardized wound closure. The experimental arm will undergo open appendectomy utilizing the Alexis® retractor, followed by standardized wound closure.
  Arms: Experimental Arm
Procedure: Open appendectomy with standardized wound closure — The control arm subjects will undergo open appendectomy and standardized wound closure. The experimental arm will undergo open appendectomy utilizing the Alexis® retractor, followed by standardized wound closure.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to determine whether the incidence of surgical site wound infection will be reduced in open appendectomy patients through the use of the Alexis® wound retractor.

DETAILED DESCRIPTION:
Aim: This is a randomized comparison of open appendectomy using metal retractors and open appendectomy using the Alexis® wound retractor in patients with simple and complicated appendicitis. The study is designed in order to minimize bias by standardizing the two procedures and blinding patients and nurses during the preoperative and postoperative period.

After obtaining informed consent, or informed assent of minors, subjects will be randomized to either of two groups: one groups will undergo a standard open appendectomy using traditional metal retractors. The second group will undergo an open appendectomy with the use of the Alexis® wound retractor.

Pre-operative antibiotic Zosyn will be given prior to skin incision. Skin prep will be betadine, duraprep or gel prep. After entering the peritoneal cavity, the Alexis® retractor will be introduced and used to maintain retraction for the duration of surgery.

In simple appendicitis, the patient will receive one dose of antibiotics six hours after surgery. The patient will not receive oral antibiotics at discharge. In complicated appendicitis, the patient will be given Zosyn until afebrile for 24 hours and a normal white blood cell count. The patient will be discharged on oral antibiotics.

Follow up will occur between the 14th and 21st post operative day. At the test of cure visit, the wound will be checked for erythema, drainage, or opening. It will be assessed whether the subject received any further medical attention or received medications since discharge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of appendicitis
* Open appendectomy
* Ability to attend follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Waxman, MD, Principal Investigator — Santa Barbara Cottage Hospital Director of Surgical Education; Todd Pederson, MD, Principal Investigator — Santa Barbara Cottage Hospital/Naval Hospital; Benedict Taylor, MD, Principal Investigator — Santa Barbara Cottage Hospital Surgical Resident; Pamela Lee, MD, Principal Investigator — Santa Barbara Cottage Hospital
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm | Control Arm
Started | 61 | 48
Completed | 61 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Control Arm | Total
Number analyzed (Participants) | 61 | 48 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (18.9) | 33.1 (16.1) | 34.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 38 | 32 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 61 | 48 | 109
Number of Participants with physical barrier to protect the wound [Count of Participants; unit: Participants] | 61 | 48 | 109

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Wound Infection, After Open Appendectomy
Description: Wound infections will be documents in both the traditional retraction arm and the wound protections device arm. The severity of appendicitis between the two groups will be matched.
Time Frame: 21 post operative days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 61 | 48
Participants | 1 | 7

ADVERSE EVENTS:
Arm/Group | Experimental Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/61 | 7/48
Other Adverse Events (participants affected / at risk) | 0/61 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=61) | Control Arm (N=48)
Wound Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7) — Wound Infection

LIMITATIONS AND CAVEATS:
This study population included gastric, hepato-biliary-pancreatic, as well as colorectal cases, whereas our study was limited to open appendectomy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No